CLINICAL TRIAL: NCT00542685
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled, Parallel Group, 10-Week Study Evaluating the Efficacy And Safety of PD 0332334 for the Treatment of Generalized Anxiety Disorder
Brief Title: A 10-Week Study Evaluating the Efficacy And Safety of PD 0332334 for the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5361017
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PD 0332334 300 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo
- PD 0332334 225 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- PD 0332334 175 mg BID (Experimental)
  Interventions: Drug: PD 0332334

INTERVENTIONS:
Drug: PD 0332334 — Capsules, oral, 300 mg BID, 8 weeks with 2 week taper.
  Other Names: imagabalin
  Arms: PD 0332334 300 mg BID
Drug: Placebo — Capsules, oral, placebo BID, 8 weeks with 2 week taper.
  Arms: Placebo BID
Drug: PD 0332334 — Capsules, oral, 225 mg BID, 8 weeks with 2 week taper.
  Arms: PD 0332334 225 mg BID
Drug: PD 0332334 — Capsules, oral, 175 mg BID, 8 weeks with 2 week taper.
  Arms: PD 0332334 175 mg BID

SUMMARY:
This study will evaluate the efficacy and safety of PD 0332334 for the treatment of generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GAD (Diagnostic and Statistical Manual-IV [DSM-IV], 300.02) as established by the clinician (psychiatrist or licensed clinical psychologist) who has interviewed the subject using all sources of data including the Mini International Neuropsychiatric Interview (MINI) for DSM-IV Axis I disorders and other clinical information. Subjects with specific phobia(s) (as defined in DSM-IV) or dysthymic disorder will be allowed in the study.
* Subjects must have a HAM-A total score ≥20 at the screening (V1) and randomization (V2) visits. Subjects must also have a Covi Anxiety Scale score of >9 and a Raskin Depression Scale score <7 at the Screening (V1) visit to ensure predominance of anxiety symptoms over depression symptoms.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, neurologic, active infections, immunological, or allergic disease (including drug allergies).
* Any of the following current (within the past 6 months through the present) DSM-IV Axis I diagnoses: Major depressive disorder, Obsessive compulsive disorder, Panic disorder; Agoraphobia, Posttraumatic stress disorder, Anorexia, Bulimia, Caffeine-induced anxiety disorder, Alcohol or substance abuse or dependence unless in full remission for at least 6 months, Social anxiety disorder.
* Any of the following past or current DSM IV Axis I diagnoses: Schizophrenia, Psychotic disorder, Delirium, dementia, amnestic, and other clinically significant cognitive disorders, Bipolar or schizoaffective disorder, Cyclothymic disorder, Dissociative disorders.
* Antisocial or borderline personality disorder.
* Serious suicidal risk per the clinical investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of PD 0332334 in the treatment of GAD will be measured by the change in the Hamilton Anxiety Rating Scale (HAM-A) total scores from baseline observed following 8 weeks of double-blind treatment. | 8 weeks
The safety and tolerability of PD 0332334 in subjects with GAD will be monitored in this study. | 8 weeks

SECONDARY OUTCOMES:
Response rate on the clinician-rated CGI-I at Week 1 and Week 8. | 8 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study-Sleep Scale (MOSS-SS) subscales. | 8 weeks
Change from Baseline to Week 8 on the Sheehan Disability Scale (SDS) total score. | 8 weeks
Change from Baseline to Days 2-8 and Weeks 2, 4, 6, 8 on the DAS-A (total score). | 8 weeks
Response rate on the HAM-A at Week 1 and Week 8. | 8 weeks
Change from Baseline in the somatic subscale score of the HAM-A (Items 7-13) at Week 8. | 8 weeks
Remission rate based on the HAM-A at Week 1 and Week 8. | 8 weeks
Response rate on the patient-rated PGI-C at Week 8. | 8 weeks
The "Week 1 Sustained Responder" rate based on the HAM-A (where "Week 1 Sustained Responders" are defined as subjects with a 50% or greater improvement from baseline on the HAM-A total score at Week 1 that is sustained until the Week 8 visit). | 1 week
Change from Baseline in HAM-A total score at Weeks 1, 2, 4, and 6. | 6 weeks
Change from Baseline in the 17-item HAM-D total score at Weeks 1, 2, 4, and 8. | 8 weeks
Change from Baseline to Week 8 on the Sheehan Disability Scale subscales. | 8 weeks
Change from Baseline in CGI-S at Week 8. | 8 weeks
Change from Baseline in the psychic subscale score of the HAM-A (Items 1-6 and 14) at Week 8. | 8 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study Sleep Scale (MOS-SS) total score. | 8 weeks
Change from Baseline to Week 8 in the Q-Les-Q General Activities Score. | 8 weeks
Change from Baseline to Week 1 on the Medical Outcomes Study Sleep Scale (MOS-SS) total score. | 1 week
Change from Baseline to Days 2-8 and Weeks 2, 4, 6, 8 on the GA-VAS (diary). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (40):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Sherman Oaks, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Lafayette, Indiana
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Belmont, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Cherry Hill, New Jersey
  - Pfizer Investigational Site, Piscataway, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Middleton, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361017&StudyName=A%2010-Week%20Study%20Evaluating%20the%20Efficacy%20And%20Safety%20of%20PD%200332334%20for%20the%20Treatment%20of%20Generalized%20Anxiety%20Disorder